CLINICAL TRIAL: NCT04425070
Title: A Phase 1/2, Open-label, Multi-center Study to Evaluate theSafety and Efficacy of Selinexor Combined With Chemotherapy orTislelizumab in Relapsed or Refractory Mature T and NK Cell Lymphoma
Brief Title: A Study of Evaluating the Safety and Efficacy of ATG-010 Combined With Chemotherapy Sequential With ATG-010 Monotherapy Maintenance in Peripheral T- and NK/T-cell Lymphoma
Acronym: TOUCH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the adjustment of clinical research and development strategy，sponsor decided to terminate the study
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-T/NK-001
Record Dates: First submitted 2020-05-25; First posted 2020-06-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T-cell Lymphoma; NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Extranodal NK-T-Cell | interventions — Ice; gemcitabine-oxaliplatin regimen; tislelizumab

STUDY DESIGN:
Intervention Model Description: ATG-010 + ICE ATG-010 + GEMOX ATG-010 + Tislelizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ATG-010 + ICE (Experimental): ATG-010 60 mg/once,total twice in each cycle; on Days 4 and 11
  Interventions: Combination Product: ICE [ifosfamide+carboplatin+etoposide]
- ATG-010 + GEMOX (Experimental): ATG-010 60 mg/once,total twice in each cycle; on Days 2 and 9
  Interventions: Combination Product: GEMOX [gemcitabine+oxaliplatin]
- ATG-010 + Tislelizumab (Experimental): ATG 010 40mg/once, will be given on Days 1, 8, and 15 of each cycle
  Interventions: Combination Product: Tislelizumab

INTERVENTIONS:
Combination Product: ICE [ifosfamide+carboplatin+etoposide] — • Combined with ICE chemotherapy regimen:
  * Ifosfamide: 5 g/m2, continuous intravenous (iv) infusion (mesna 5 g/m2 synchronously iv infusion for rescue), on Day 2;
  * Carboplatin: with concentration-area under time curve (AUC)=5 (highest concentration to 800 mg), iv infusion, on Day 2;
  * Etoposide l00 mg/m2, iv infusion, on Days 1-3;
  * ATG-010 60 mg/once, oral, on Days 4 and 11. After the treatment with combination chemotherapy, the patients will continue to receive maintenance treatment of ATG-010 60 mg/once per week (QW).
  Arms: ATG-010 + ICE
Combination Product: GEMOX [gemcitabine+oxaliplatin] — • Combined with GEMOX chemotherapy regimen:
  * Gemcitabine 1000 mg/m2, iv infusion, on Days 1 and 8;
  * Oxaliplatin 130 mg/m2, iv infusion, on Day 1;
  * ATG-010 60 mg/once, oral, on Days 2 and 9. After the treatment with combination chemotherapy, the patients will continue to receive maintenance treatment of ATG-010 60 mg/once per week (QW).
  Arms: ATG-010 + GEMOX
Combination Product: Tislelizumab — Tislelizumab will be administered intravenously at a fixed dose of 2 0 0 mg every 3 weeks on Day 1 of each cycle
  Arms: ATG-010 + Tislelizumab

SUMMARY:
This trial is proposed with treatment of ATG-010 combined with chemotherapy regimens which will be chosen by investigators (ICE [ifosfamide+carboplatin+etoposide] or GEMOX [gemcitabine+oxaliplatin] or Tislelizumab), after treatments of 2 to 6 cycles transferring to ATG-010 monotherapy maintenance treatment, to evaluate the safety, tolerability, and primary efficacy of ATG-010 in R/R PTCL and NK/T-cell lymphoma patients.

DETAILED DESCRIPTION:
This trial is an open-label, multi-center Phase Ib clinical study that will evaluate ATG-010 combined with chemotherapy regimen selected by investigators (ICE regimen ifosfamide+carboplatin+etoposide; Or GEMOX regimen: gemcitabine+oxaliplatin; Tislelizumab) sequential ATG 010 monotherapy maintenance, to evaluate the safety, tolerability, and primary efficacy in R/R PTCL and NK/T-cell lymphoma patients. 97 patients are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing to provide written ICF.
2. Age≥ 18 years.
3. R/R PTCL and NK/T-cell lymphoma as confirmed by histological methods according to WHO classification of tumors of lymphoid tissues 2016.
4. Previously received at least one or more standard regimens including anthracycline.
5. Recurrence or the recurrence disease after the last treatment completed.
6. At least one measurable disease per modified efficacy assessment criteria (Cheson 2014).
7. ECOG PS 0 or 1.
8. Any toxicity caused by previously anti-tumor therapy must recovered to ≤ Grade 1 (NCI-CTCAE v5.0) with exception of hearing loss, alopecia, and pigmentation.
9. Expected life time longer than 3 months.

Exclusion Criteria:

1. Current have disease or history of central nervous system lymphoma.
2. HBV-DNA positive, or HCV-RNA positive.
3. Patients with a known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.
4. Received major surgery within 4 weeks of first dose of study drug
5. Known received SINE, including ATG-010.
6. Unable to swallow the tablets, suffers from malabsorption syndrome, or any other gastrointestinal disease or dysfunction that may interfere with ATG-010 absorption.
7. Known allergy to ATG-010, or ICE, or GEMOX.
8. A woman who is pregnant or nursing.
9. The investigator considerations on patient's complications or other conditions may affect protocol compliance or may be inappropriate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
AEs/SAEs | 18 months
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.
Overall Response Rate (ORR) | 18 months
  To determine the overall response rate according to Chenson 2014.

SECONDARY OUTCOMES:
Duration of response (DOR) | 18 months
  Duration of time from first occurrence of CR or PR until the first date that disease progression is objectively documented.
Disease control rate (DCR) | 4 weeks to 18 months
  Proportion of patients who achieve CR, PR, or SD for a minimum of 4 weeks, following the first dose of study drug (i.e., CR+PR+SD)
Progression-free survival (PFS) | 18 months
  Duration of time from the first dose of study drug until progression or death due to any cause
Overall Survival (OS) | 18 months
  Duration of time from the first dose of study drug until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yu, MD, Study Director — Medical Director
Locations (13):
- China (13):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Tongren Hospital.CMU, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical Universisity Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang